CLINICAL TRIAL: NCT01296503
Title: Thalidomide Plus Dexamethasone as Maintenance Therapy After Autologous Hematopoietic Stem Cell Transplantation for Multiple Myeloma: a Multicenter Phase 3 Randomized Trial
Brief Title: Thalidomide Plus Dexamethasone as Maintenance Therapy for Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo de Estudos Multicentricos em Onco-Hematologia (Network)
Responsible Party: Angelo Maiolino, MD, PhD, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBRAM0001
Record Dates: First submitted 2011-01-27; First posted 2011-02-15 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Treatment; Maintenance; Thalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Arm A) (Active Comparator): Sixty days (D+60) after ASCT: randomization in two arms of maintenance: Arm A (dexamethasone alone 40 mg/day for 4 days every 28 days)
  Interventions: Drug: Dexamethasone
- Thalidomide and Dexamethasone (Arm B) (Experimental): D+60 after ASCT: dexamethasone plus thalidomide 200 mg by mouth daily for 12 months or until disease progression.
  The dose of thalidomide could be reduced if the patient experienced grade 2 or higher adverse events. In this case, thalidomide was discontinued and re-challenged at a lower dose after resolution of the adverse event.
  Interventions: Drug: Thalidomide plus dexamethasone

INTERVENTIONS:
Drug: Thalidomide plus dexamethasone — D+60 after ASCT: randomization in two arms of maintenance: Arm A (dexamethasone alone 40 mg/day for 4 days every 28 days) and Arm B (dexamethasone plus thalidomide 200 mg by mouth daily) for 12 months or until disease progression.
  The dose of thalidomide could be reduced if the patient experienced grade 2 or higher adverse events. In this case, thalidomide was discontinued and re-challenged at a lower dose after resolution of the adverse event.
  Other Names: Thalomid; Baycadron; DexPak; Decadron
  Arms: Thalidomide and Dexamethasone (Arm B)
Drug: Dexamethasone — dexamethasone alone 40 mg/day for 4 days every 28 days
  Other Names: Baycadron; DexPak; Decadron
  Arms: Dexamethasone (Arm A)

SUMMARY:
This multicenter, prospective, randomized trial was designed to evaluate the role of thalidomide with or without dexamethasone as a maintenance therapy for multiple myeloma patients after a single autologous stem cell transplantation.

DETAILED DESCRIPTION:
Patients were recruited prior to receiving induction therapy, and randomization in a 1:1 ratio occurred on day 60 post-autologous stem cell transplantation. The treatment consisted of the following four phases:

1. induction with 3-5 cycles of vincristine plus doxorrubicin and dexamethasone (VAD) every 21-28 days: vincristine 0.4 mg , doxorubicin 9 mg/m² and oral dexamethasone 40 mg daily for 4 days;
2. cyclophosphamide (4 g/m2 ) plus filgrastim (G-CSF) (5 μg/kg twice a day) for stem cell mobilization;
3. melphalan (200 mg/m2 ) and one autologous stem cell transplant (ASCT);
4. Sixty days (D +60) after ASCT: RANDOMIZATION in two arms of maintenance: Arm A (oral dexamethasone alone 40 mg/d for 4 days every 28 days) and Arm B (dexamethasone plus thalidomide 200 mg daily by mouth) for 12 months or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic multiple myeloma in accordance with the International Myeloma Working Group criteria;
* age 18-70 years;
* Performance status 0-2 by the Eastern Cooperative Oncology Group (ECOG) criteria;
* normal hepatic function, defined as serum bilirubin <3 mg/dl and alanine aminotransferase(ALT) and asparagin aminotransferase (AST) <4x normal.

Exclusion Criteria:

* evidence of disease progression after ASCT;
* cardiac dysfunction (systolic ejection fraction <50%);
* chronic respiratory disease (carbon monoxide diffusion <50% of normal).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2003-10; Primary Completion 2008-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Progression Free survival | 36 months
  Primary endpoint: progression free survival (PFS) PFS was defined as the time between randomization and any documentation of relapse, progression, or death by any cause.

SECONDARY OUTCOMES:
Overall survival | 36 months
  Secondary endpoints: overall survival (OS) was defined as the interval from randomization to death (or the last follow-up for surviving patients). For patients who were not randomized, OS was calculated from the date of diagnosis until the date of death or last follow-up.
safety of thalidomide | 36 months
  The number of patients experiencing adverse events grade 3 or 4 were compared between treatment arms. Adverse events were classified as defined by the National Cancer Institute Common Toxicity Criteria, version 2. Safety evaluations were focused especially on neurological symptoms and the development of deep venous thrombosis (DVT). Adverse events evaluations were performed at the time of response assessment and whenever a new clinical manifestation suggestive of toxicity appeared.

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Maiolino, MD, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (4):
- Brazil (4):
  - Hospital Universitário Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro
  - Universidade Estadual de Campinas, Campinas, São Paulo
  - Universidade de São Paulo- Ribeirão Preto, Ribeirão Preto, São Paulo
  - Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo